CLINICAL TRIAL: NCT01643837
Title: Mastalgia Treatment: Is There a Role for Osteopathic Manipulative Treatment?
Brief Title: Mastalgia Treatment: Is There a Role for Osteopathic Manipulative Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to free investigators; time constraints
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BHS-799
Record Dates: First submitted 2012-07-10; First posted 2012-07-18 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Mastalgia
Keywords: Mastalgia; Breast Pain; Osteopathic Manipulative Medicine; Osteopathic Manipulative Treatment
MeSH Terms: conditions — Mastodynia | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard (No Intervention): Standard treatment follow-up: 1. monthly history 2. monthly clinical breast examination.
- Light Touch (LT) (Sham Comparator): Standard treatment follow-up: 1. monthly history 2. monthly clinical breast examination.
  Light touch protocol.
  Interventions: Other: Osteopathic Manipulative Light Touch Protocol (LT)
- Osteopathic Manipulative Treatment (OMT) (Experimental): Standard treatment follow-up: 1. monthly history 2. monthly clinical breast examination.
  OMT Protocol.
  Interventions: Other: Osteopathic Manipulative Treatment

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment — OMT - Sacral Ligamenotus Articular Release; OMT - Lumbar Spine (L1-L2) and Lower Thoracic Spine (T10-12) Ligamentous Articular Release; OMT - Upper Thoracic Spine Ligamentous Articular Release (T1-T8); OMT - Cervical Spine Ligamentous Articular Release (C5-C7); OMT - Suboccipital Myofascial Release; OMT - Clavicular Ligamentous Articular Release; OMT - First Rib Ligamentous Articular Release; OMT - Ribs 2-8 Ligamentous Articular Release; OMT - Pectoral Pull; OMT - Sternal Ligamentous Articular Release; OMT - Direct Myofascial Release of the Diaphragm; OMT - Thoracic Lymphatic Pump; OMT - Fascial Release of Breast Tissue
  Arms: Osteopathic Manipulative Treatment (OMT)
Other: Osteopathic Manipulative Light Touch Protocol (LT) — LT - Sacral Region; LT - Lumbar Spine and Lower Thoracic Region; LT - Upper Thoracic Spine Region; LT - Cervical Spine Region; LT - Suboccipital Region; LT - Clavicles; LT - First Ribs; LT - Ribs 2-8; LT - Pectoralis Muscles; LT - Sternum; LT - Respiratory Diaphragm; LT - Upper Thoracic Cage; LT - Lower Thoracic Cage
  Arms: Light Touch (LT)

SUMMARY:
There are many current medical treatments for mastalgia, but few have been proven effective. Our objective is to evaluate the effectiveness of osteopathic manipulative treatment as compared to a light touch protocol and standard management in the treatment of women with cyclical and non-cyclical mastalgia. We will compare duration of the pain, severity of the pain and the effect of the pain on quality of life.

DETAILED DESCRIPTION:
Our objective is to evaluate the effectiveness of osteopathic manipulative treatment (OMT) as compared to a light touch protocol and standard management in the treatment of women with cyclical and non-cyclical mastalgia (breast pain).

A randomized placebo controlled study will be conducted at two academic health care centers. Women with breast pain will be evaluated and followed by the breast surgeon. Once a pathologic cause has been ruled out, the women will be stratified and randomly divided into three study groups. Group A, B, and C. Group A will receive standard of care treatment. Group B will receive light touch (a placebo for the OMT treatment). Group C will receive OMT directed at treating mastalgia. The treatment will continue for three months.

The subjects will fill out an initial pain questionnaire and a follow-up questionnaire each month. They will also be instructed to fill out a breast pain log daily for three months. A final questionnaire will be completed at six months. Statistical analysis will be utilized to determine whether the addition of OMT improves the severity or duration of the pain as well as quality of life as assessed by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age presenting with breast pain, both cyclical and noncyclical, who complain of pain despite a negative full work-up for pathology, reassurance, and use of an appropriate supportive bra.
* A pain scale questionnaire will be completed by the subject. The pain should be present for at least 7 days each month if it is mild pain or be of moderate to severe intensity for at least 3 days each month. In addition, breast pain must have been present for a minimum of 2 consecutive months preceding the date of inclusion into the study.

Exclusion Criteria:

* Women under 18 years old, women who have had recent breast surgery (<2yrs), women who have breast implants.
* Women with bleeding risk such as those regularly taking aspirin, NSAIDs, Plavix or any other anticoagulation therapy.
* Women who are pregnant, breastfeeding or who are planning to get pregnant are excluded.
* Women with known chronic pain syndromes or structural abnormality such as osteoporosis will be excluded. When necessary bone densitometry will be performed.
* Women who are unable to complete the questionnaire.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Severity of Mastalgia | 30, 60, 90, 120, 210 days
Change from baseline in Duration of Mastalgia | 30, 60, 90, 120, 210 days
Change from baseline in Quality of Life | 30, 60, 90, 120, 210 days

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Koehler, DO, Principal Investigator — New York Institute of Technology
Locations (2):
- United States (2):
  - Family Health Care Center, Central Islip, New York
  - Academic Health Care Center, Old Westbury, New York

REFERENCES:
- [Background] Khan SA, Apkarian AV. The characteristics of cyclical and non-cyclical mastalgia: a prospective study using a modified McGill Pain Questionnaire. Breast Cancer Res Treat. 2002 Sep;75(2):147-57. doi: 10.1023/a:1019685829799. PMID 12243507
- [Background] Rosolowich V, Saettler E, Szuck B; BREAST DISEASE COMMITTEE. RETIRED: Mastalgia. J Obstet Gynaecol Can. 2006 Jan;28(1):49-57. doi: 10.1016/S1701-2163(16)32027-8. English, French. PMID 16533457
- [Background] Ader DN, Browne MW. Prevalence and impact of cyclic mastalgia in a United States clinic-based sample. Am J Obstet Gynecol. 1997 Jul;177(1):126-32. doi: 10.1016/s0002-9378(97)70450-2. PMID 9240595
- [Background] Nichols S, Waters WE, Wheeler MJ. Management of female breast disease by Southampton general practitioners. Br Med J. 1980 Nov 29;281(6253):1450-3. doi: 10.1136/bmj.281.6253.1450. PMID 7437833
- [Background] Hughes LE, Mansel RE, Webster DJT. Breast pain and nodularity. Benign Disorders and Diseases of the Breast. London, England: Saunders 2000:95-121.
- [Background] Millet AV, Dirbas FM. Clinical management of breast pain: a review. Obstet Gynecol Surv. 2002 Jul;57(7):451-61. doi: 10.1097/00006254-200207000-00022. PMID 12172222
- [Background] Srivastava A, Mansel RE, Arvind N, Prasad K, Dhar A, Chabra A. Evidence-based management of Mastalgia: a meta-analysis of randomised trials. Breast. 2007 Oct;16(5):503-12. doi: 10.1016/j.breast.2007.03.003. Epub 2007 May 16. PMID 17509880
- [Background] Pain JA, Cahill CJ. Management of cyclical mastalgia. Br J Clin Pract. 1990 Nov;44(11):454-6. PMID 2282296
- [Background] Still AT. Osteopathy research and practice. Seattle, WA: Eastland Press; 1992.
- [Background] Andersson GB, Lucente T, Davis AM, Kappler RE, Lipton JA, Leurgans S. A comparison of osteopathic spinal manipulation with standard care for patients with low back pain. N Engl J Med. 1999 Nov 4;341(19):1426-31. doi: 10.1056/NEJM199911043411903. PMID 10547405
- [Background] Kuchera W, Kuchera M. Osteopathic principles in practice. 2nd ed. Dayton, OH: Greyden Press; 1994.
- [Background] Chila AG, et al. Foundations for osteopathic medicine. 3rd ed. Philadelphia, PA: Lippincott Williams and Wilkins; 2011.
- [Background] Nelson KE. Somatic dysfunction in osteopathic family medicine. 2nd ed. Baltimore, MD: Lippincott Williams & Wilkins; 2007.
- [Background] Kuchera W, Kuchera M. Osteopathic Considerations in Systemic Dysfunction. revised 2nd ed. Dayton, OH: Greyden Press; 1994.
- [Background] ACS guidelines http://www.cancer.org/Healthy/FindCancerEarly/CancerScreening Guidelines/american-cancer-society-guidelines-for-the-early-detection-of-cancer. Accessed 5.14.11.
- [Background] DiGiovanna EL, Schiowitz S, editors. An osteopathic approach to diagnosis and treatment. 2nd ed. Philadelphia, PA: Lippincott-Raven Publishers; 1997.